CLINICAL TRIAL: NCT01820195
Title: The Effect of N-Acetyl Cystein in Preventing Contrast Induced Nephropathy: A Double Blind Double Dummy Randomized Controlled Trial
Brief Title: N-Acetyl Cystein and Contrast Nephropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Khomeini Hospital (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Principal Investigator, Mohammad Reza Khatami, Associate professor, Imam Khomeini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: THC-18043
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease Stage 2; Radiographic Contrast Agent Nephropathy
Keywords: Contrast Nephropathy; N-Acetyl Cystein; Prophylaxy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous N Acetyl Cystein (Active Comparator): 1200 mg IV N- Acetyl Cystein half an hour before contrast administration. This group will also take oral placebo
  Interventions: Drug: IV N-Acetyl Cystein
- Placebo (Placebo Comparator): Patients on both oral placebo and IV placebo just like patients on oral and IV N-acetyl cystein groups in regard of dose and timing.
  Interventions: Drug: Placebo group
- Oral N Acetyl Cystein (Active Comparator): Patients on 600 mg oral N-Acetyl Cystein bid started at the day before contrast exposure and continue until the next day of contrast exposure.These patients will also take IV placebo
  Interventions: Drug: Oral N-Acetyl Cystein

INTERVENTIONS:
Drug: Oral N-Acetyl Cystein — Oral N-Acetyl Cystein 600 mg bid started the day before contrast administration and continue the day after exposure to contrast
  Arms: Oral N Acetyl Cystein
Drug: IV N-Acetyl Cystein — Bolus IV administration of 1200 mg N- Acetyl Cystein half an hour before contrast media administration
  Arms: Intravenous N Acetyl Cystein
Drug: Placebo group — The patients in this group will be received both oral placebo and IV placebo
  Arms: Placebo

SUMMARY:
There are many controversies about the role of N-Acetyl Cystein in preventing of contrast nephropathy. These contradictory results may be due to different criteria for patients' selection, different end points, different type and dose of N-Acetyl Cystein administration and finally different prophylactic measures other than N-Acetyl Cystein. The investigators try to enroll a double blind double dummy study with a good power to compare the effect of this drug both in the form of oral and intravenous against the placebo in preventing the contrast nephropathy in the patients whom undergo coronary angiography/angioplasty.

DETAILED DESCRIPTION:
Contrast Nephropathy is the third cause of acute kidney injury in hospitalized patients. The morbidity and mortality of this disorder is considerable. There is no treatment for this condition and all measures should be taken into account to prevent this complication. Among the all prophylactic measures hydration and the dose ant type of contrast are the only factors that have been proved to be effective in preventing contrast nephropathy. N-Acetyl Cystein is an antioxidant agents that may be effective in different aspects of medicine, but it,s use in this condition is controversial. While some studies showed it is effective in prevention of contrast nephropathy, others showed no benefit. Different studies used different dose and route of administration. So more clinical trials with good power are needed to compare different oral Vs IV administration of the drug in a randomized double blinded clinical trial. In this study we allocate the eligible patients with chronic kidney diseases stages 2 to 4 to three groups. Oral N-Acetyl Cystein group, IV N-Acetyl Cystein group, placebo group. All group will be matched according to stages of chronic kidney diseases, diabetes, anemia, heart failure, age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* chronic Kidney disease stage 2-4
* use of nephrotoxins in last week leading to angiography

Exclusion Criteria:

* Acute kidney injury
* concomitant use of other nephrotoxins
* need of repeated imaging with contrast in five days after the first surgery
* need for surgery in next five day after the contrast exposure
* need of using nephrotoxins in next five days after contrast exposure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Increase in serum creatinine more than 25% of baseline | 24 hours, 48 hours after exposure to contrast media

SECONDARY OUTCOMES:
Increase in serum creatinine more than 25% of baseline | The 5th day after exposure to contrast media

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Khatami, MD, Study Chair — Nephrology Research Center; Ebrahin Kassaian, MD, Principal Investigator — Tehran Heart Center; Mojtaba Salarifar, MD, Principal Investigator — Tehran Heart Center; Ali Kazemi-Saeid, MD, Principal Investigator — Tehran Heart Center
Locations (1):
- Tehran Heart Center, Tehran, Iran